CLINICAL TRIAL: NCT04517942
Title: An Evaluation of the Peer-delivered EVERYbody Project: Eating Disorder Risk Factor Reduction for College Students
Brief Title: Evaluation of Peer-led EVERYbody Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Washington University (Other)
Responsible Party: Principal Investigator, Anna Ciao, Associate Professor of Psychology, Western Washington University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 17-004_2
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Body Image; Eating Disorder Symptom
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: After signing up for a specific time slot, participants were randomized in blocks of 10 to the EVERYbody Project or video comparison condition (two blocks of 10 participant slots were available in each time slot).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVERYbody Project: Peer facilitator version (Experimental): This dissonance-based body image program was created from focus group feedback (Ciao, Ohls, & Pringle, 2017) and piloted in an initial randomized-controlled trial. Based on the Body Project (Stice et al., 2006), it retains key dissonance activities while adapting exercises to have a more inclusive focus (e.g., expanding the gender focus, exploring diversity characteristics within appearance ideals, adjusting activities to be inclusive of diversity).
  Around 10% of the original EVERYbody Project manual was modified to create the Peer Facilitator version for the current trial. Changes focused on adding individual exercises to draw out the critique of diversity in cultural ideals, refining prompts to be more suitable for peer facilitation, and flagging sections of the manual for more "expert" peer facilitation.
  Peer facilitators received 16 hours of training on the EVERYbody Project manual and peer facilitation guidelines (e.g., group management, handling problems, etc.).
  Interventions: Behavioral: EVERYbody Project
- Video + Expressive Writing group (Active Comparator): Video + expressive writing groups were facilitated by a peer leader following a detailed script. This intervention was designed as an active but low-dissonance comparison condition. Participants viewed two separate documentary movies related to gender and/or appearance-related pressures (one during each session): (1) The Illusionists (2015 ), and (2) The Mask You Live In (2015). Participants engaged in a brief (10 minute) reflective writing exercise after each film. In order to keep dissonance low, participants were told that their reflections would not be shared with anyone and they were not turned in.
  Peer facilitators received brief (1 hour) training on the video group manual.
  Interventions: Other: Video + Expressive Writing

INTERVENTIONS:
Behavioral: EVERYbody Project — Brief behavioral intervention (4 hours across two meetings)
  Arms: EVERYbody Project: Peer facilitator version
Other: Video + Expressive Writing — Brief video-based intervention (4 hours across two meetings)
  Arms: Video + Expressive Writing group

SUMMARY:
The second trial of the EVERYbody Project explored the efficacy of the inclusive body image intervention when delivered by college peer leaders. The peer-facilitated EVERYbody Project was compared to a video and expressive writing comparison intervention through one-month follow-up.

DETAILED DESCRIPTION:
The initial trial of the EVERYbody Project established that professional leaders could deliver a universal, inclusive body image program for college students, with benefit above and beyond a waitlist control condition. The second trial of the EVERYbody Project aimed to further evaluate the intervention using a more disseminable facilitator model: trained college student peer leaders. It also utilized a more rigorous comparison condition, where peer leaders conducted the two-session EVERYbody Project program or a time-matched video and expressive writing intervention. College students within a university in the Pacific Northwest United States were invited to participate in programming (universal intervention target). Quantitative assessment included a comparison of changes in eating disorder risk factor outcomes across randomization conditions at pre- and post-intervention and one-month follow-up. Feasibility and acceptability explored the impact of the peer delivered program within universal college student audiences.

ELIGIBILITY:
Inclusion Criteria:

* Current college student enrolled at institution where research was taking place

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Eating disorder symptoms | Assessed at baseline (Survey 1), post-intervention (Survey 2), and one-month follow-up (Survey 3)
  Eating disorder symptoms were assessed with the Eating Disorders Examination Questionnaire (EDEQ; Fairburn & Beglin, 1994). The Global score of the EDEQ was used in this study (average across all 28 items).
Body dissatisfaction | Assessed at baseline (Survey 1), post-intervention (Survey 2), and one-month follow-up (Survey 3)
  The Satisfaction and Dissatisfaction with Body Parts Scale (SDBPS; Berscheid, Walster, & Bohrnstedt, 1973) assessed satisfaction and dissatisfaction with nine parts of the body that are commonly endorsed as concerning (e.g., stomach, thighs, hips). The average score was used in this study (average across all 9 items).
Internalized cultural appearance norms | Assessed at baseline (Survey 1), following intervention Session 1 (Survey 1.B), post-intervention (Survey 2), and one-month follow-up (Survey 3)
  The two Internalization subscales of the Sociocultural Attitudes Toward Appearance Questionnaire-4 (SATAQ-4; Schaefer et al., 2015) assess internalized cultural messages surrounding appearance and attractiveness. The two internalization subscales were combined for this study (average across all 10 items), following prior research by Kilpela et al. (2016). This survey was assessed at all outcome time points (Survey 1, 2, and 3), plus midway through the intervention (following Session 1 of the program).

SECONDARY OUTCOMES:
Negative affect | Assessed at baseline (Survey 1), post-intervention (Survey 2), and one-month follow-up (Survey 3)
  Negative affect was assessed with 20 items from the fear, guilt, and sadness subscales of the Positive and Negative Affect Schedule-Revised (PANAS-X; Watson & Clark, 1992). The average of all 20 items was used in this study.

OTHER OUTCOMES:
Program satisfaction and application | Assessed at post-intervention (Survey 2) and one-month follow-up (Survey 3).
  A series of feedback questions were used to gauge satisfaction with the EVERYbody Project (based on Ciao et al., 2015). These questions included four Likert scale items about enjoyment (e.g., "I enjoyed the EVERYbody Project") rated from 1 (strongly disagree) to 5 (strongly agree) as well as open-ended questions (e.g., "Was any part of the EVERYbody Project particularly helpful/useful? If so, which part and why?") These questions were administered immediately following participation in the EVERYbody Project as a part of the post-intervention survey (Survey 2).
  At post-intervention (Survey 2) and one-month follow-up (Survey 3), three questions gauged application of information learned in the program (e.g., "How often do think about the things you learned in the EVERYbody Project?" rated on a scale from 1 (not at all) to 5 (all the time).

CONTACTS AND LOCATIONS:
Overall Officials: Anna C Ciao, PhD, Principal Investigator — Western Washington University
Locations (1):
- Western Washington University, Bellingham, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and other materials will be made available following reasonable request to study Principal Investigator. All outcome data will be included in data sharing. Socio-demographic characteristics will be collapsed into broader categories to protect participant identity.
  Other study materials, including intervention manuals, will be housed on the Principal Investigator's Open Science Framework page, where URLs will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Since the trial is complete, data are available immediately upon request.
URL: https://osf.io/x3k7v/?view_only=c9dbd31a4ad94a08b16421d719bc0fac

REFERENCES:
- [Background] Ciao AC, Ohls OC, Pringle KD. Should body image programs be inclusive? A focus group study of college students. Int J Eat Disord. 2018 Jan;51(1):82-86. doi: 10.1002/eat.22794. Epub 2017 Nov 6. PMID 29105805
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Schaefer LM, Burke NL, Thompson JK, Dedrick RF, Heinberg LJ, Calogero RM, Bardone-Cone AM, Higgins MK, Frederick DA, Kelly M, Anderson DA, Schaumberg K, Nerini A, Stefanile C, Dittmar H, Clark E, Adams Z, Macwana S, Klump KL, Vercellone AC, Paxton SJ, Swami V. Development and validation of the Sociocultural Attitudes Towards Appearance Questionnaire-4 (SATAQ-4). Psychol Assess. 2015 Mar;27(1):54-67. doi: 10.1037/a0037917. Epub 2014 Oct 6. PMID 25285718
- [Background] Stice E, Shaw H, Burton E, Wade E. Dissonance and healthy weight eating disorder prevention programs: a randomized efficacy trial. J Consult Clin Psychol. 2006 Apr;74(2):263-75. doi: 10.1037/0022-006X.74.2.263. PMID 16649871
- [Background] Berscheid, E., Hatfield [Walster], E., & Bohrnstedt, G. (1973). The happy American body: A survey report. Psychology Today, 7, 119-131.
- [Background] Watson, D., & Clark, L. A. (1992). Affects separable and inseparable: On the hierarchical arrangement of the negative affects. Journal of Personality and Social Psychology, 62, 489-505. http://dx.doi.org/10.1037/ 0022-3514.62.3.489
- [Background] Ciao AC, Latner JD, Brown KE, Ebneter DS, Becker CB. Effectiveness of a peer-delivered dissonance-based program in reducing eating disorder risk factors in high school girls. Int J Eat Disord. 2015 Sep;48(6):779-84. doi: 10.1002/eat.22418. Epub 2015 May 8. PMID 25959408
- [Background] Kilpela LS, Blomquist K, Verzijl C, Wilfred S, Beyl R, Becker CB. The body project 4 all: A pilot randomized controlled trial of a mixed-gender dissonance-based body image program. Int J Eat Disord. 2016 Jun;49(6):591-602. doi: 10.1002/eat.22562. Epub 2016 May 18. PMID 27188688
- [Result] Ciao AC, Munson BR, Pringle KD, Roberts SR, Lalgee IA, Lawley KA, Brewster J. Inclusive dissonance-based body image interventions for college students: Two randomized-controlled trials of the EVERYbody Project. J Consult Clin Psychol. 2021 Apr;89(4):301-315. doi: 10.1037/ccp0000636. PMID 34014692